CLINICAL TRIAL: NCT00740727
Title: Enzymatically Augmented Subcutaneous Infusion (EASI) Access II Trial
Brief Title: EASI Access II --- Follow-up Study to the EASI Access Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Stephen H. Thomas MD MPH, Massachusetts General Hospital/Harvard Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EASI Access II
Record Dates: First submitted 2008-08-21; First posted 2008-08-25 (Estimated); Results first posted 2009-09-11 (Estimated); Last update posted 2009-09-11 (Estimated); Status verified 2009-09

CONDITIONS: Disaster Medicine; Difficult Intravenous Access; Dehydration
Keywords: Disaster; Mass casualty incident; Prehospital; Rehydration; Intravascular access
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EASI (Experimental): Subjects will undergo placement of EASI catheters. All subjects in whom EASI catheters are placed, will receive Human Recombinant Hyaluronidase (HRH) as part of the EASI placement. (No subject will receive HRH, other than as part of EASI catheter placement.)
  Interventions: Drug: Human recombinant hyaluronidase (HRH); Procedure: Enzymatically Augmented Subcutaneous Infusion (EASI) line placement

INTERVENTIONS:
Drug: Human recombinant hyaluronidase (HRH) — 150u HRH administered via EASI access line, prior to infusion of 250 D5W (5% dextrose in water)
  Other Names: Hylenex
Procedure: Enzymatically Augmented Subcutaneous Infusion (EASI) line placement — Subjects will under placement of an EASI line. This entails placement of a small (20-gauge) catheter in the upper back, in the subcutaneous space.

SUMMARY:
Test whether Basic Life Support (BLS) providers can successfully place Enzymatically Augmented Subcutaneous Infusion (EASI) Access lines for subcutaneous infusion, and characterize intravascular absorption of EASI-administered (tracer-labelled) glucose (D5W).

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be at least 18 years of age and have none of the following conditions:

  * pregnancy (negative urine pregnancy test to be performed before study participation),
  * diabetes, or coagulopathic (including taking any anticoagulants);
* Subjects cannot be taking steroids or other immunosuppressants.
* Because of the potential for reduced hyaluronidase effectiveness, the study excludes patients taking more than 80 mg daily aspirin, as well as any patients taking ACTH, antihistamines, or estrogen other than in oral contraceptive preparations.
* Subjects will not be required to fast before the study, but will not allowed to eat or drink during the EASI infusion or the phlebotomy sampling time frame.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen H Thomas, MD MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Sever MS, Vanholder R, Lameire N. Management of crush-related injuries after disasters. N Engl J Med. 2006 Mar 9;354(10):1052-63. doi: 10.1056/NEJMra054329. No abstract available. PMID 16525142
- [Background] Stafford PW, Blinman TA, Nance ML. Practical points in evaluation and resuscitation of the injured child. Surg Clin North Am. 2002 Apr;82(2):273-301. doi: 10.1016/s0039-6109(02)00006-3. PMID 12113366
- [Background] Bookbinder LH, Hofer A, Haller MF, Zepeda ML, Keller GA, Lim JE, Edgington TS, Shepard HM, Patton JS, Frost GI. A recombinant human enzyme for enhanced interstitial transport of therapeutics. J Control Release. 2006 Aug 28;114(2):230-41. doi: 10.1016/j.jconrel.2006.05.027. Epub 2006 Jun 7. PMID 16876899
- [Background] Thomas JR, Yocum RC, Haller MF, von Gunten CF. Assessing the role of human recombinant hyaluronidase in gravity-driven subcutaneous hydration: the INFUSE-LR study. J Palliat Med. 2007 Dec;10(6):1312-20. doi: 10.1089/jpm.2007.0126. PMID 18095810
- [Background] Beylot M, David F, Brunengraber H. Determination of the 13C-labeling pattern of glutamate by gas chromatography-mass spectrometry. Anal Biochem. 1993 Aug 1;212(2):532-6. doi: 10.1006/abio.1993.1364. PMID 8105720
- [Background] Bijur PE, Latimer CT, Gallagher EJ. Validation of a verbally administered numerical rating scale of acute pain for use in the emergency department. Acad Emerg Med. 2003 Apr;10(4):390-2. doi: 10.1111/j.1553-2712.2003.tb01355.x. PMID 12670856
- [Background] Alam HB, Rhee P. New developments in fluid resuscitation. Surg Clin North Am. 2007 Feb;87(1):55-72, vi. doi: 10.1016/j.suc.2006.09.015. PMID 17127123
- [Background] Dalal S, Bruera E. Dehydration in cancer patients: to treat or not to treat. J Support Oncol. 2004 Nov-Dec;2(6):467-79, 483. PMID 15605914
- [Background] Craig AS, Eikenberry EF, Parry DA. Ultrastructural organization of skin: classification on the basis of mechanical role. Connect Tissue Res. 1987;16(3):213-23. doi: 10.3109/03008208709006977. PMID 2956050
- [Background] Laurent UB, Dahl LB, Reed RK. Catabolism of hyaluronan in rabbit skin takes place locally, in lymph nodes and liver. Exp Physiol. 1991 Sep;76(5):695-703. doi: 10.1113/expphysiol.1991.sp003536. PMID 1742011
- [Background] Frost GI. Recombinant human hyaluronidase (rHuPH20): an enabling platform for subcutaneous drug and fluid administration. Expert Opin Drug Deliv. 2007 Jul;4(4):427-40. doi: 10.1517/17425247.4.4.427. PMID 17683255
- [Derived] Soremekun OA, Shear ML, Connolly J, Stewart CE, Thomas SH. Basic-level emergency medical technician administration of fluids and glucose via enzyme-assisted subcutaneous infusion access. Prehosp Disaster Med. 2012 Jun;27(3):220-5. doi: 10.1017/S1049023X12000829. PMID 22854002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred in January 2009
Pre-assignment Details: A total of 20 subjects were consented. The study day ran long, so 2 subjects who had consented (and had an initial intravenous {IV} access placed, but no EASI access placed) declined to have any of the study procedures performed since the 2-hour phlebotomy window would have kept them at the study site until the evening.
Groups:
- EASI/HRH(Human Recombinant Hyaluronidase): Subjects underwent placement of EASI (Enzymatically Augmented Subcutaneous Infusion) catheters
Period: Overall Study
Arm/Group | EASI/HRH(Human Recombinant Hyaluronidase)
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | EASI/HRH(Human Recombinant Hyaluronidase)
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successfully Placed EASI Lines
Description: Ability of Basic Life Support (BLS) providers to place EASI access lines.
  The unit of analysis is the 18 BLS participants (these were also the 18 individuals in whom the EASI access lines were placed).
Time Frame: 1 day
Population: Participants received EASI access placement, with co-administration of human recombinant hyaluronidase.
Measure: Number; unit: Participants
Arm/Group | EASI/HRH(Human Recombinant Hyaluronidase)
Number analyzed (Participants) | 18
Participants | 18

2. Primary Outcome: Systemic Absorption of Subcutaneously Administered Tracer-labelled Glucose
Description: Number of subjects (out of a possible 18) in whom EASI-administered tracer-labeled glucose was absorbed systemically.Gas chromatography/Mass spectrometry analysis was performed on timed phlebotomy samples, to assess for tracer-labeled glucose.Isotopic glucose enrichment was determined by plasma analysis on a Hewlett-Packard 5985B quadruple mass spectrometer, using + chemical ionization (methane reagent gas). A 12m×0.20mm ID, OV-1 capillary column (He carrier) was used in the gas chromatograph.Enrichments of glucose were calculated as atom percent excess relative to natural background level.
Time Frame: 1 day
Population: Participants received EASI access placement, with co-administration of human recombinant hyaluronidase.
Measure: Number; unit: Participants
Arm/Group | EASI/HRH(Human Recombinant Hyaluronidase)
Number analyzed (Participants) | 18
Participants | 18

3. Secondary Outcome: Number of Participants With Pain During EASI Infusion
Description: Assessment during EASI placement & initial infusion, for pain as assessed with 10-point scale (0=no pain; 10=worst pain). Significant pain was defined a priori as a pain score of at least 3.
Time Frame: 1 day
Population: Participants received EASI access placement, with co-administration of human recombinant hyaluronidase.
Measure: Number; unit: Participants
Arm/Group | EASI/HRH(Human Recombinant Hyaluronidase)
Number analyzed (Participants) | 18
Participants | 2
Statistical Analysis 1: Comparison: EASI/HRH(Human Recombinant Hyaluronidase); This analysis reports the number of subjects (of 18 possible) who experienced pain, during EASI placement or infusion, at the a priori-defined level of at least 3 on a 10-point pain scale; Test type: Superiority or Other; 95% binomial exact confidence interval; % of subjects with infusion pain = 11.1, 95% CI [1.4 to 34.7]

4. Secondary Outcome: Number of Participants With Pain at EASI Infusion Site, on Next-day Follow-up
Description: Assessment during upon next-day follow-up, for pain as assessed with 10-point scale (0=no pain; 10=worst pain). Significant pain was defined a priori as a pain score of at least 3.
  Presence of any pain (yes or no question and then numeric rating if pain was present) was assessed upon follow-up by telephone; on this follow-up a yes/no question was also asked about any complications at infusion site (in the upper back).
Time Frame: 2 days
Population: Participants received EASI access placement, with co-administration of human recombinant hyaluronidase.
Measure: Number; unit: Participants
Arm/Group | EASI/HRH(Human Recombinant Hyaluronidase)
Number analyzed (Participants) | 18
Participants | 0
Statistical Analysis 1: Comparison: EASI/HRH(Human Recombinant Hyaluronidase); This analysis reports the number of subjects (of 18 possible) who experienced pain, as assessed on next-day follow-up (24 hours after EASI infusion), at the a priori-defined level of at least 3 on a 10-point pain scale; Test type: Superiority or Other; binomial exact confidence interval; Because the point estimate was zero, the statistical software (STATA version 10MP) reports a one-sided 97.5% confidence interval; % subjects with next-day EASI site pain = 0, 97.5% CI [0 to 18.5]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No